CLINICAL TRIAL: NCT02357056
Title: Randomized Controlled Evaluation of Robotic Cardiac Surgery Training Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 106343
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Robotic Surgery Simulation Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wet Lab (Active Comparator): Subjects in the wet lab group will perform dissections of the internal thoracic artery and placement of annuloplasty stitches in the mitral valve in pig models until time proficiency is reached based on the performance of our expert robotic surgeons.
  Interventions: Other: Wet Lab
- Dry Lab (Active Comparator): Subjects in the dry lab group will perform exercises form the fundamentals of laparoscopic surgery (FLS) program adapted for the daVinci robot. These exercises included, camera and clutching, peg transfer and intracorporeal knot tying. Participants will repeat these tasks until time proficiency is reached based on the performance of our expert robotic surgeons.
  Interventions: Other: Dry Lab
- Virtual Reality (Active Comparator): Subjects in the virtual reality group will perform exercises from a 9 task curriculum, on the daVinci Skills Simulator. These exercises included, camera and clutching, energy switching, peg board, energy dissection, matchboard, ringwalk, suture sponge, and vertical defect suturing. Participants will repeat these tasks all metrics are passed and an overall score is reached based on the performance of our expert robotic surgeons.
  Interventions: Other: Virtual Reality
- Control (No Intervention): The control group will receive no training after they complete the initial assessment and undergo randomization. They will be invited back after several weeks to complete the final assessment to control for any improvement in performance from the initial assessment alone and normal progression through surgical training outside of this project.

INTERVENTIONS:
Other: Wet Lab — ITA dissection and Annuloplasty Sutures in porcine model.
  Arms: Wet Lab
Other: Dry Lab — Camera and clutching, peg transferring, intracorporeal knot tying
  Arms: Dry Lab
Other: Virtual Reality — daVinci Surgical Skills simulation
  Arms: Virtual Reality

SUMMARY:
The purpose of this research is to objectively compare various training modalities currently available in minimally invasive and robotic surgery to determine the most effective training methods specific to robotic cardiac surgery. We hope to recruit medical trainees with minimal robotic surgery training experience, randomly assigned to one of three groups (Dry wab, da Vinci Simulator and Wet lab). Trainees will be evaluated at baseline for a standardized tasks common in robotic cardiac surgery and then divided into one of the three training modalities. Trainees will be given sufficient time to become proficient with a variety of predetermined tasks unique to each training group. The trainees will then undergo a reevaluation with the cardiac surgery specific tasks at the end of a standard training period. We will then be able to compare our three groups to show if any have benefits over the others in regards to improvement in technical ability, understanding of the robots functions, efficacy of training, speed of technical skill development, accuracy and efficiency of movement. We will rate each modality on their reproducibility, accuracy of representation, and ease of set up and perform a cost analysis for each of the training methods.

ELIGIBILITY:
Inclusion Criteria:

* Residents, fellows and staff of a surgical specialty with less then 10 hours using the daVinci robot or any robotic simulator.

Exclusion Criteria:

* Individuals not associated with a surgical program
* Individuals with >10 hours experience driving the daVinci Robot or any robotic simulator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Time to Complete Mitral Valve Annuloplasty | 3 months
  A total score for this task will be generated from the formula; Score = 720 - Time(s), If any damage is done to the tissues a score of zero will be assessed.
Time To Complete 10cm dissection of the Internal Thoracic Artery | 3 months
  A total score for this task will be generated from the formula; Score = 1320 - Time(s), If any damage is done to the tissues a score of zero will be assessed.
Global Evaluative Assessment of Robotic Skills (GEARS) Score | 3 Months
  A validated objective scoring tool will be used to evaluate overall robotic surgical skill for each task.

SECONDARY OUTCOMES:
Duration of Training | 3 Months
  Total duration of time spent on the robot in order to reach proficiency marks set by expert surgeons will be recorded and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Bob Kiaii, MD, Principal Investigator — Department of Cardiac Surgery
Locations (1):
- Canadian Surgical Technologies & Advanced Robotics (CSTAR), London, Ontario, Canada

REFERENCES:
- [Derived] Valdis M, Chu MW, Schlachta CM, Kiaii B. Validation of a Novel Virtual Reality Training Curriculum for Robotic Cardiac Surgery: A Randomized Trial. Innovations (Phila). 2015 Nov-Dec;10(6):383-8. doi: 10.1097/IMI.0000000000000222. PMID 26680752